CLINICAL TRIAL: NCT04760197
Title: ASIA Study: French Register of Inflammatory Eye Disease Secondary to Cancer Immunotherapy
Brief Title: ASIA Study : French Register of Inflammatory Eye Disease
Acronym: ASIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_0136
Record Dates: First submitted 2021-02-16; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Patients Treated for Cancer by Immunotherapy
Keywords: immune check points" inhibitors; cancer; inflammatory ophthalmological manifestations
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patient under cancer immunotherapy with inflammatory ophthalmological manifestations: patient(>18 years old) under cancer immunotherapy with inflammatory ophthalmological manifestations
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
New anticancer therapies based on lifting the inhibition of the immunological synapse are used in the therapeutic arsenal of a growing number of neoplasias (melanoma, lung cancer, hepatocellular carcinoma, etc.). These "immune check points" inhibitors "(ICPI) target molecules that usually allow immunity to destroy malignant cells. At the systemic level, this results in a loss of immune homeostasis and facilitation of the inflammatory response which may be responsible for dysimmune manifestations distant from the neoplastic site. Thus, since their introduction, ICPIs have been of interest to immunologists, rheumatologists and internists who often find themselves in the first line to deal with this type of side effect (immunotherapy-related adverse events, IRAEs). The frequency of these ARIs between 70% and 90%, depending on the immunotherapy used and the severity of these ARIIs (grade 1-2 vs. 3-5). The overall increase in the number of cancers, the multiplication of available molecules and the expansion of their indications should exponentially increase the number of IRAEs to be supported. Little is known about the epidemiology, risk factors and efficacy of treatments.

In these IRAEs, inflammatory ophthalmological manifestations have been described with an estimated prevalence of between 0.4 and 1% of the patients treated. These attacks are rare and protean (uveitis, scleritis, retinitis, inflammatory orbitopathies, Vogt-Koyanagi-Harada -like…) and reported most often in the form of clinical cases.

The Main objective is to describe the inflammatory ophthalmic disorders linked to anti-cancer immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* age> 18
* under cancer immunotherapy: anti-PD1 (nivolumab, pembrolizumab), anti-CTLA4 (ipilimumab), anti-PDL1 (atezolizumab, durvalumab, avelumab)
* diagnosis of uveitis / inflammatory ophthalmologic disease confirmed by at least an ophthalmologist
* indicating his/her non-opposition to participating in the study

Exclusion Criteria:

* NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients treated for cancer by immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Clinical evolution of inflammatory ophtalmological manifestation evaluated by gradation of uveitis | 6 months after diagnosis
  Persistence of disease is characterized by persistence of intraocular inflammation evaluated by gradation of Uveitis according to Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0, November 2017, National Institutes of Health, National Cancer Institute.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Chaudot, MD, Principal Investigator — : Hospices Civils de Lyon - Groupement Hospitalier Nord
Locations (2):
- France (2):
  - CHU Angers - Service de Médecine Interne - Immunologie Clinique, Angers
  - Hôpital de la Croix-Rousse - Service de médecine interne - 103 Grande Rue de la Croix-Rousse, Lyon